CLINICAL TRIAL: NCT07356219
Title: The Merits of the Prognostic Nutritional Index for Prediction of the Outcome of Coronary Artery Bypass Grafting Surgery: A Retrospective Observational Study
Brief Title: Prognostic Nutritional Index for Predicting Outcomes Following Coronary Artery Bypass Grafting (CABG) Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohammed El Gazzar, Assistant professor of Cardiothoracic Surgery, Faculty of Medicine, Benha University, Egypt, Benha University
Other Study IDs: RC 6.11.2025
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Body Mass Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABG Patient Cohort.: Patients who underwent Coronary Artery Bypass Grafting surgery at Benha University Hospital over the preceding five years.
  Interventions: Diagnostic Test: Prognostic Nutritional Index (PNI); Diagnostic Test: Neutrophil-to-Lymphocyte Ratio (NLR); Diagnostic Test: Body Mass Index (BMI)

INTERVENTIONS:
Diagnostic Test: Prognostic Nutritional Index (PNI) — Calculated using serum albumin (g/L) and total peripheral lymphocyte count.
Diagnostic Test: Neutrophil-to-Lymphocyte Ratio (NLR) — Calculated from peripheral blood counts.
Diagnostic Test: Body Mass Index (BMI) — Calculated from preoperative weight and height.

SUMMARY:
Coronary artery bypass grafting (CABG) is a major cardiac surgery associated with risks of serious perioperative complications and mortality. Malnutrition and inflammation are known independent risk factors for poor outcomes in patients with coronary artery disease. This retrospective observational study evaluates the Prognostic Nutritional Index (PNI)-a simple score derived from serum albumin and lymphocyte counts-as an objective measure of nutritional and inflammatory status. The research aims to determine how well preoperative PNI and its postoperative changes can predict complications such as acute kidney injury, myocardial infarction, and sternal wound infections in patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent CABG surgery.
* Availability of a signed informed consent form before surgery.

Exclusion Criteria:

* Other concurrent cardiac surgeries.
* Presence of malignancy or systemic inflammatory disorders.
* Active infection or autoimmune disorders.
* Maintenance on immunosuppressants.
* Liver disease.
* Files with missing data.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of adult patients (both male and female) who underwent major coronary artery bypass grafting surgery at the Cardiothoracic Surgery Department of Benha University Hospital within a recent five-year period.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-01-11 (Actual); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the Prognostic Nutritional Index (PNI) in Predicting Post-CABG Complications. | Approximately 30 days (From surgery through the duration of the hospital/ICU stay.)
  The Area Under the Receiver Operating Characteristic (ROC) Curve (AUC) used to determine the performance of the PNI score in predicting the occurrence of major postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Al Qalyoubia, Egypt